CLINICAL TRIAL: NCT04941170
Title: U/s Guided Oblique Subcostal Transversus Abdominis Plane Block Versus Erector Spinae Plane Block as Pre-emptive Analgesia for Open Umbilical Hernia Repair; Randomized, Double-blinded Controlled Trial
Brief Title: U/s Guided Oblique Subcostal Transversus Abdominis Plane Block Versus Erector Spinae Plane Block as Preemptive Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Abdel Fatah, Lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC 2-6-2021
Record Dates: First submitted 2021-06-19; First posted 2021-06-28 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Pain; Hernia, Umbilical
Keywords: Open umbilical hernia; Transversus abdominis plane block; Erector spinae plane block
MeSH Terms: conditions — Pain; Hernia, Umbilical | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (T) (Active Comparator): receive preoperative bilateral ultrasound-guided oblique subcostal transversus abdominis plane block.
  Interventions: Drug: Bupivacain; Drug: Bupivacaine
- Group (E) (Active Comparator): receive preoperative bilateral ultrasound-guided erector spinae plane block.
  Interventions: Drug: Bupivacain; Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacain — Ultrasound-guided oblique subcostal transversus abdominis plane block will be performed in the supine position under strict aseptic precautions. placing a linear high-frequency ultrasound probe obliquely near the costal margin and xiphoid process On confirming the placement of the needle in the correct target space, 1 mL of 0.25% bupivacaine will be injected to hydro-dissect the fascia layer between the RA and TA. After confirming the separation of the transversus abdominis fascia plane, the remaining 19 mL of 0.25% bupivacaine will be administered, advancing the needle infero-laterally parallel to the subcostal margin. A similar procedure will be performed on the contralateral side of the abdomen with an injection of another 20 mL of 0.25% bupivacaine.
  Other Names: oblique subcostal transversus abdominis plane block
Drug: Bupivacaine — Ultrasound-guided erector spinae plane block will be performed in the sitting position. T7 spinous process will be located To perform the block. The tip of the T7 transverse process will be then identified using the ultrasound probe that is placed in a transverse orientation The ultrasound transducer will then be placed in a longitudinal orientation 2-3 cm lateral to the midline in a longitudinal orientation to identify the hyperechoic line of the transverse process with its associated acoustic shadow. After local anaesthetic infiltration, the block needle will be inserted in a craniocaudal direction until contact will be achieved with the T 7 transverse process where the tip will lay in the inter-fascial plane below the erector spinae muscle. A small bolus of local anaesthetic should be given through the block needle to confirm the proper needle position. A total of 20 mL bupivacaine 0.25% will be injected into the interfacial plane deep to the erector spinae muscle bilaterally.
  Other Names: erector spinae plane block

SUMMARY:
Administration of opioids for the treatment of acute pain after open umbilical hernia repair is associated with many side effects. Erector spinae plane (ESP) block is a novel inter-fascial plane block used in postoperative pain and chronic neuropathic pain relief of the thoracoabdominal region.TAP block is a regional injection of local anaesthetic between the transversus abdominis and internal oblique muscle planes. TAP block affects the sensory nerves of the anterolateral abdominal wall (T6-L1) that innervate the abdomen.

DETAILED DESCRIPTION:
TAP block is a regional injection of local anaesthetic between the transversus abdominis and internal oblique muscle planes. TAP block affects the sensory nerves of the anterolateral abdominal wall (T6-L1) that innervate the abdomen. TAP block is an easy technique and decreases postoperative pain and opioid consumption.

Erector spinae plane (ESP) block is a novel inter-fascial plane block used in postoperative pain and chronic neuropathic pain relief of the thoracoabdominal region. However, its first use was for the treatment of chronic pain, but recently it has been used as a postoperative regional analgesia technique in different surgeries from the shoulder to hip regions (3-4) The present study will be carried out to compare the preemptive analgesic efficacy between the ultrasound-guided bilateral ESP block versus bilateral oblique subcostal TAP block on patients undergoing open umbilical hernia repair.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of anesthesiologists I-II, scheduled for open umbilical hernia repair.
2. Age range of 18-65 years.

Exclusion Criteria:

1. patient refusal.
2. Patients belonging to ASA grade III and grade IV.
3. Extreme obesity (BMI >35).
4. hepatic or renal insufficiency.
5. preoperative cognitive dysfunction or communication disorder.
6. allergy to amide-type local anaesthetics.
7. back puncture site infection.
8. Coagulation disorders, pregnancy, drug abusers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
total morphine consumption. | in first 24 hours
  Amount of morphine used as rescue analgesia post-operatively.

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | From the start of operation till its end up to 3 hours.
  Intraoperative fentanyl dosage (μg)
time of first analgesic request | in 24 hours
  first time of analgesia used after operation.
pain severity evaluation. | at PACU admission , 30 minutes , 2 hours , 4 hours , 8 hours ,12 hours ,18 hours and 24 hours post operative
  by verbal numerical rating scale (VNRS) at rest and cough (0 = no pain, 10 = unbearable pain).

CONTACTS AND LOCATIONS:
Overall Officials: fatma ah abdelfatah, MD, Principal Investigator — Benha University
Locations (1):
- Banha Faculity of Medicine, Banhā, Elqalyoubea, Egypt